CLINICAL TRIAL: NCT02745080
Title: A Randomized, Double-blind, Active Control, Multicenter Study to Evaluate the Efficacy at Week 52 of Secukinumab Monotherapy Compared With Adalimumab Monotherapy in Patients With Active Psoriatic Arthritis
Brief Title: Efficacy of Secukinumab Compared to Adalimumab in Patients With Psoriatic Arthritis
Acronym: EXCEED 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2366; 2015-004477-32 (EudraCT Number)
Record Dates: First submitted 2016-04-01; First posted 2016-04-20 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; secukinumab; adalimumab; monoclonal antibody; CASPAR
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Secukinumab 300 mg s.c. (Experimental): Secukinumab 300 mg administered at Baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks until Week 48.
  Interventions: Biological: Secukinumab
- Adalimumab 40 mg s.c. (Active Comparator): Adalimumab 40 mg administered at Baseline followed by dosing every 2 weeks until Week 50.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Secukinumab — Eligible subjects are randomized to one of two treatment arms in a 1:1 ratio
  Other Names: AIN457
  Arms: Secukinumab 300 mg s.c.
Biological: Adalimumab — Eligible subjects are randomized to one of two treatment arms in a 1:1 ratio
  Arms: Adalimumab 40 mg s.c.

SUMMARY:
This was a randomized, double-blind, active controlled, multicenter, parallel-group study evaluating secukinumab monotherapy and adalimumab monotherapy in approximately 850 patients with active psoriatic arthritis (PsA) who are naïve to biologic therapy and are intolerant or having inadequate response to conventional disease modifying anti-rheumatic drugs (also known as non-biologic DMARDs).

DETAILED DESCRIPTION:
The total maximum study duration, including the screening period was up to 76 weeks.

At Baseline, patients whose eligibility was confirmed were randomized to 1 of 2 groups (1:1): Group 1 (secukinumab 300 mg) or Group 2 (adalimumab 40 mg).

In order to maintain the blind, both groups received 1 or 2 placebo s.c. injections to keep consistency in the number of injections at each dosing visit. Secukinumab (300 mg) was available in 2 x 1.0 mL pre-filled syringes (PFS) and adalimumab was available in 1 x 0.4 mL PFS. Placebo (1.0 and 0.5 mL PFS) was also available.

Secukinumab 300 mg s.c injection (2 x 1 mL PFS) was administered at Baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks to Week 48.

Adalimumab 40 mg (1 x 0.4 mL PFS) was administered at Baseline followed by dosing every 2 weeks until Week 50.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of PsA classified by CASPAR
* Rheumatoid factor and anti-CCP antibodies negative
* Diagnosis of active plaque psoriasis, with at least one psoriatic plaque of >= 2cm diameter or nail changes consistent with psoriasis or documented history of plaque psoriasis
* Inadequate control of symptoms with NSAIDs
* Inadequate control of symptoms with a conventional DMARD.

Key Exclusion Criteria:

* Pregnant or nursing women
* Evidence of ongoing infectious or malignant process
* Previous exposure to any biologic drug for Psoriatic Arthritis or Psoriasis
* Subjects taking high potency opioid analgesics
* Ongoing use of prohibited psoriasis treatments/medications
* Previous treatment with any cell-depleting therapies including but not limited to anti-CD20 investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (137):
- United States (19):
  - Novartis Investigative Site, Fountain Valley, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, La Mesa, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Bethlehem, Pennsylvania
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Arlington, Texas
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Glendale, Wisconsin
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern East, Victoria
- Bulgaria (3):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (3):
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (4):
  - Novartis Investigative Site, Bruntál
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
  - Novartis Investigative Site, Zlín
- Novartis Investigative Site, Frederiksberg, Denmark
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Finland (2):
  - Novartis Investigative Site, Hyvinkää
  - Novartis Investigative Site, Kuopio
- France (7):
  - Novartis Investigative Site, Brive-la-Gaillarde
  - Novartis Investigative Site, Cahors
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Poitiers
- Germany (10):
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Schwerin
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Veszprém
- Novartis Investigative Site, Reykjavik, Iceland
- India (4):
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Secunderabad, Telangana
  - Novartis Investigative Site, New Delhi
- Israel (5):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (6):
  - Novartis Investigative Site, Arenzano, GE
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Torino
- Latvia (2):
  - Novartis Investigative Site, Riga
  - Novartis Investigative Site, Valmiera
- Lithuania (3):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda
  - Novartis Investigative Site, Šiauliai
- Netherlands (2):
  - Novartis Investigative Site, Enschede
  - Novartis Investigative Site, Sneek
- Poland (3):
  - Novartis Investigative Site, Dopiewo
  - Novartis Investigative Site, Szczecin
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Ponte de Lima
  - Novartis Investigative Site, Porto
- Russia (8):
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Nizhny Novgorod
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (4):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Partizánske
  - Novartis Investigative Site, Topoľčany
- Novartis Investigative Site, Seoul, Seocho Gu, South Korea
- Spain (19):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Mérida, Extremadura
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- United Kingdom (14):
  - Novartis Investigative Site, Torquay, Devon
  - Novartis Investigative Site, Leytonstone, London
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Cannock, Staffordshire
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Solihull
  - Novartis Investigative Site, Wigan
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Kaeley GS, Schett G, Conaghan PG, McGonagle D, Behrens F, Goupille P, Gaillez C, Parikh B, Bakewell C. Enthesitis in patients with psoriatic arthritis treated with secukinumab or adalimumab: a post hoc analysis of the EXCEED study. Rheumatology (Oxford). 2024 Jan 4;63(1):41-49. doi: 10.1093/rheumatology/kead181. PMID 37097894
- [Derived] McInnes IB, Behrens F, Mease PJ, Kavanaugh A, Ritchlin C, Nash P, Masmitja JG, Goupille P, Korotaeva T, Gottlieb AB, Martin R, Ding K, Pellet P, Mpofu S, Pricop L; EXCEED Study Group. Secukinumab versus adalimumab for treatment of active psoriatic arthritis (EXCEED): a double-blind, parallel-group, randomised, active-controlled, phase 3b trial. Lancet. 2020 May 9;395(10235):1496-1505. doi: 10.1016/S0140-6736(20)30564-X. PMID 32386593
- See also: Secukinumab versus adalimumab for treatment of active psoriatic arthritis (EXCEED): a double-blind, parallel-group, randomised, active-controlled, phase 3b trial — https://pubmed.ncbi.nlm.nih.gov/32386593/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 161 centers in 26 countries worldwide: Australia, Bulgaria, Canada, Czech Republic, Denmark, Estonia, Finland, France, Germany, Greece, Hungary, Iceland, India, Israel, Italy, South Korea, Latvia, Lithuania, The Netherlands, Poland, Portugal, Russia, Slovakia, Spain, UK and USA.
Pre-assignment Details: 853 patients were randomized in a 1:1 ratio to receive secukinumab 300 mg (N=426) or adalimumab 40 mg (N=427); All randomized patients were analyzed for efficacy and safety.
Period: Overall Study
Arm/Group | Secukinumab 300 mg s.c. | Adalimumab 40 mg s.c.
Started (All randomized patients were included in the Full Analysis Set (FAS) and Safety Analysis Set (SAF)) | 426 | 427
Completed | 371 | 338
Not Completed | 55 | 89
Not completed — Adverse Event | 13 | 21
Not completed — Lack of Efficacy | 11 | 23
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 3 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 22 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg s.c. | Adalimumab 40 mg s.c. | Total
Number analyzed (Participants) | 426 | 427 | 853
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.5 (12.38) | 49.5 (12.44) | 49.0 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 198 | 416
  Male | 208 | 229 | 437
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 16 | 20 | 36
  American Indian or Alaska Native | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 402 | 391 | 793
  Unknown | 1 | 5 | 6
  Other | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 20% (ACR20) Response at Week 52
Description: Clinical response, failure to permanently discontinue study medication prematurely, and lack of need for rescue medication was required for a patient to achieve treatment success. The primary endpoint is the proportion of patients with monotherapy ACR20 response at Week 52 where monotherapy ACR20 response is defined as meeting the following 3 conditions:
  1. achieving American College of Rheumatology 20 (ACR20) response
  2. no permanent study treatment (secukinumab or adalimumab) discontinuation before or at Week 50 (the last dosing visit)
  3. no use of conventional disease modifying anti-rheumatic drugs (also known as non-biologic DMARDs) cDMARDs (including Methotrexate (MTX)) after Week 36 (regardless of the starting time of taking cDMARDs)
Time Frame: Week 52
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Secukinumab 300 mg s.c. | Adalimumab 40 mg s.c.
Number analyzed (Participants) | 426 | 427
Percentage of Participants | 67.4 [62.8 to 71.7] | 61.5 [56.8 to 66.0]
Statistical Analysis 1: Comparison: Secukinumab 300 mg s.c. vs Adalimumab 40 mg s.c; Test type: Superiority; p = 0.0719, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.98 to 1.72] — Odds ratio, 95% confidence interval, and p-value are from a logistic regression model with treatment as a factor and baseline weight as a covariate

2. Secondary Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index (PASI)-90 Response at Week 52
Description: The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Time Frame: Week 52
Population: Psoriasis Subset of the Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Secukinumab 300 mg s.c. | Adalimumab 40 mg s.c.
Number analyzed (Participants) | 215 | 202
Percentage of Participants | 65.4 [58.8 to 71.5] | 43.2 [36.5 to 50.2]
Statistical Analysis 1: Comparison: Secukinumab 300 mg s.c. vs Adalimumab 40 mg s.c; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.49, 95% CI 2-sided [1.67 to 3.71] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology 50% (ACR50) Response at Week 52
Description: Clinical response, failure to permanently discontinue study medication prematurely, and lack of need for rescue medication was required for a patient to achieve treatment success. The secondary endpoint is the proportion of patients with monotherapy ACR50 response at Week 52 where monotherapy ACR50 response is defined as meeting the following 3 conditions:
  1. achieving American College of Rheumatology 50 (ACR50) response
  2. no permanent study treatment (secukinumab or adalimumab) discontinuation before or at Week 52
  3. no use of conventional disease modifying anti-rheumatic drugs (also known as non-biologic DMARDs) cDMARDs (including Methotrexate (MTX)) after Week 36 (regardless of the starting time of taking cDMARDs)
Time Frame: Week 52
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Secukinumab 300 mg s.c. | Adalimumab 40 mg s.c.
Number analyzed (Participants) | 426 | 427
Percentage of Participants | 49.0 [44.3 to 53.7] | 44.8 [40.1 to 49.5]
Statistical Analysis 1: Comparison: Secukinumab 300 mg s.c. vs Adalimumab 40 mg s.c; Test type: Superiority; p = 0.2251, Regression, Logistic; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.90 to 1.55] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI Score) at Week 52
Description: The HAQ-DI assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 52
Population: Full Analysis Set (FAS)
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Secukinumab 300 mg s.c. | Adalimumab 40 mg s.c.
Number analyzed (Participants) | 426 | 427
Unit on a scale | -0.58 (0.027) | -0.56 (0.027)
Statistical Analysis 1: Comparison: Secukinumab 300 mg s.c. vs Adalimumab 40 mg s.c; Test type: Superiority; p = 0.5465, Mixed Models Analysis; least squares (LS) mean change = -0.02, 95% CI 2-sided [-0.10 to 0.05], Standard Error of Mean 0.038 — Mixed model repeated measures (MMRM) with treatment group, analysis visit as factors, weight/baseline score as covariates, treatment by analysis visit, baseline score by analysis visit as interation terms and unstructured covariance structure

5. Secondary Outcome: Percentage of Participants Who Achieved Resolution of Enthesitis at Week 52
Description: Enthesitis refers to inflammation of entheses, the site where ligaments or tendons insert into the bones. Resolution was defined as the absence of recorded enthesitis; conducted by the study assessor.
Time Frame: Week 52
Population: Enthesitis Subset (LEI) of the Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Secukinumab 300 mg s.c. | Adalimumab 40 mg s.c.
Number analyzed (Participants) | 234 | 264
Percentage of Participants | 60.5 [54.1 to 66.6] | 54.2 [48.2 to 60.2]
Statistical Analysis 1: Comparison: Secukinumab 300 mg s.c. vs Adalimumab 40 mg s.c; Test type: Superiority; p = 0.1498, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.91 to 1.87] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from first dose of study treatment until 12 Weeks (84 days) following the last administration of study treatment, an average of 68 weeks.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post-treatment.
Groups:
- AIN457 300 mg: Secukinumab 300 mg administered at Baseline, Weeks 1, 2, 3 and 4, followed by dosing every 4 weeks until Week 48.
- Adalimumab 40 mg: Adalimumab 40 mg administered at Baseline followed by dosing every 2 weeks until Week 50.
- Total: Total
Arm/Group | AIN457 300 mg | Adalimumab 40 mg | Total
All-Cause Mortality (participants affected / at risk) | 1/426 | 0/427 | 1/853
Serious Adverse Events (participants affected / at risk) | 37/426 | 36/427 | 73/853
Other Adverse Events (participants affected / at risk) | 226/426 | 236/427 | 462/853
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=426) | Adalimumab 40 mg (N=427) | Total (N=853)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 1
Splenic artery aneurysm (Gastrointestinal disorders) | 0 | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Bursitis infective (Infections and infestations) | 0 | 1 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 1 | 0 | 1
Measles (Infections and infestations) | 0 | 1 | 1
Mycobacterial infection (Infections and infestations) | 0 | 1 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 3 | 3
Puncture site abscess (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Varicella (Infections and infestations) | 1 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
VIIIth nerve injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Horner's syndrome (Nervous system disorders) | 0 | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Radiculopathy (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 2 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 2
Prostatitis (Reproductive system and breast disorders) | 0 | 2 | 2
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AIN457 300 mg (N=426) | Adalimumab 40 mg (N=427) | Total (N=853)
Diarrhoea (Gastrointestinal disorders) | 32 | 37 | 69
Injection site reaction (General disorders) | 4 | 28 | 32
Bronchitis (Infections and infestations) | 16 | 27 | 43
Nasopharyngitis (Infections and infestations) | 88 | 84 | 172
Upper respiratory tract infection (Infections and infestations) | 42 | 54 | 96
Arthralgia (Musculoskeletal and connective tissue disorders) | 29 | 31 | 60
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 31 | 48
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 34 | 38 | 72
Headache (Nervous system disorders) | 36 | 33 | 69
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 14 | 38
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 25 | 15 | 40
Psoriasis (Skin and subcutaneous tissue disorders) | 33 | 34 | 67
Hypertension (Vascular disorders) | 27 | 24 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-24): https://cdn.clinicaltrials.gov/large-docs/80/NCT02745080/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02745080/SAP_001.pdf